CLINICAL TRIAL: NCT06980805
Title: A Phase 2b, Randomized, Double-blind, Placebo-controlled Study to Assess the Safety, Tolerability, and Efficacy of IMVT-1402 in Participants With Active Subacute Cutaneous Lupus Erythematosus (SCLE) and/or Chronic Cutaneous Lupus Erythematosus (CCLE) With or Without Systemic Manifestations
Brief Title: A Study to Assess the Safety, Tolerability, and Efficacy of IMVT-1402 in Participants With Cutaneous Lupus Erythematosus (CLE)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Immunovant Sciences GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IMVT-1402-2701
Record Dates: First submitted 2025-05-08; First posted 2025-05-20 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Subacute Cutaneous Lupus Erythematosus; Chronic Cutaneous Lupus Erythematosus
Keywords: Chronic Cutaneous Lupus Erythematosus; Subacute Cutaneous Lupus Erythematosus; IMVT-1402
MeSH Terms: conditions — Lupus Erythematosus, Cutaneous; Lupus Erythematosus, Discoid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Period 1: Placebo (Placebo Comparator): Matching placebo for 12 weeks in Period 1
  Interventions: Drug: Placebo
- IMVT-1402 Subcutaneous (SC) Once weekly (QW) (Experimental): * Period 1: IMVT-1402 Dose 1 SC QW for 12 weeks
  * Period 2: IMVT-1402 Dose 1 SC QW for 14 weeks
  * Period 3: IMVT-1402 Dose 1 or Dose 2 SC QW for 26 weeks
  Interventions: Drug: IMVT-1402

INTERVENTIONS:
Drug: IMVT-1402 — Dose 1 or Dose 2 SC QW
  Arms: IMVT-1402 Subcutaneous (SC) Once weekly (QW)
Drug: Placebo — Matching Placebo SC QW
  Arms: Period 1: Placebo

SUMMARY:
The primary purpose of this study is to evaluate the efficacy, safety, and tolerability of IMVT-1402 in participants with Cutaneous Lupus Erythematosus.

The study will consist of 3 periods:

Period 1: eligible participants will be randomized 1:1 to IMVT-1402 Dose 1 or placebo SC QW for 12 weeks.

Period 2: participants who completed Period 1 will receive IMVT-1402 Dose 1 SC QW for 14 weeks.

Period 3: after completion of Period 2, participants will be re-randomized 1:1 to blinded IMVT-1402 Dose 1 or Dose 2 SC QW for 26 weeks.

DETAILED DESCRIPTION:
The total study duration per participant is approximately 61 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have documented diagnosis of SCLE or CCLE that has been confirmed by biopsy with or without systemic LE manifestations.
* Have a total CLASI-A score of ≥10 at Screening and Day 1. Participants with a CLASI-A score of ≥8 and <10 are eligible if the score does not include alopecia and/or mucous membrane lesions.
* Have active CLE despite an adequate trial of conventional therapies.
* Are positive for at least one autoantibody at Screening.

Exclusion Criteria:

* Have known or suspected drug-induced CLE anti-phospholipid disease, or neuropsychiatric SLE.
* Have rapidly progressive nephritis.
* Have current inflammatory skin disease other than SCLE/CCLE that, in the opinion of the Investigator, could interfere with the inflammatory skin assessments or confound the disease activity assessments.

Note: Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-02-19 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Percent change from Period 1 Baseline in Cutaneous Lupus Erythematosus Disease area and Severity Index activity (CLASI-A) score at Week 12 | Baseline (Day 1) and Week 12
  The CLASI-A score represents the overall severity of cutaneous lupus erythematosus (CLE) dermatologic involvement. It is used to assess the activity of mucocutaneous lesions in patients with lupus. The score ranges from 0 (no active lesions) to a maximum of 70. Values between 1 and 9 indicate mild inflammation, 10 to 20 indicate moderate inflammation, and 21 or higher indicate severe inflammation.

SECONDARY OUTCOMES:
Proportion of participants who have a reduction in CLASI-A score of ≥ 5 points from Period 1 Baseline at Week 12 | Baseline (Day 1) and Week 12
Proportion of participants who have a reduction in CLASI-A score of ≥ 50% from Period 1 Baseline at Week 12 | Baseline (Day 1) and Week 12
Proportion of participants who have a reduction in CLASI-A score of ≥ 70% from Period 1 Baseline at Week 12 | Baseline (Day 1) and Week 12

CONTACTS AND LOCATIONS:
Locations (82):
- United States (32):
  - Site Number - 1010, Anniston, Alabama
  - Site Number - 1020, Birmingham, Alabama
  - Site Number - 1038, Phoenix, Arizona
  - Site Number - 1034, Scottsdale, Arizona
  - Site Number - 1022, Beverly Hills, California
  - Site Number - 1018, Chula Vista, California
  - Site Number - 1005, Fremont, California
  - Site Number - 1023, Los Angeles, California
  - Site Number - 1000, Aurora, Colorado
  - Site Number - 1033, Castle Rock, Colorado
  - Site Number - 1021, Farmington, Connecticut
  - Site Number - 1014, Hialeah, Florida
  - Site Number - 1017, Jacksonville, Florida
  - Site Number - 1028, Miami, Florida
  - Site Number - 1024, Miami, Florida
  - Site Number - 1027, Miami, Florida
  - Site Number - 1011, Miami Lakes, Florida
  - Site Number - 1025, Orlando, Florida
  - Site Number - 1009, Buford, Georgia
  - Site Number - 1030, Brighton, Massachusetts
  - Site Number - 1019, Auburn Hills, Michigan
  - Site Number - 1003, Saint Clair Shores, Michigan
  - Site Number - 1013, Troy, Michigan
  - Site Number - 1004, Saint Joseph, Missouri
  - Site Number - 1026, St Louis, Missouri
  - Site Number - 1007, Charlotte, North Carolina
  - Site Number - 1008, Durham, North Carolina
  - Site Number - 1006, Smithfield, North Carolina
  - Site Number - 1002, Hershey, Pennsylvania
  - Site Number - 1015, Philadelphia, Pennsylvania
  - Site Number - 1035, Houston, Texas
  - Site Number - 1012, Irving, Texas
- Argentina (5):
  - Site Number -5004, CABA
  - Site Number - 5000, CABA
  - Site Number - 5001, CABA
  - Site Number - 5002, San Miguel de Tucumán
  - Site Number - 5003, San Miguel de Tucumán
- Bulgaria (5):
  - Site Number - 5601, Sofia
  - Site Number - 5603, Sofia
  - Site Number - 5600, Sofia
  - Site Number - 5605, Sofia
  - Site Number - 5606, Sofia
- Chile (5):
  - Site Number - 5702, Independencia
  - Site Number - 5704, Santiago
  - Site Number - 5703, Santiago
  - Site Number - 5701, Temuco
  - Site Number - 5700, Victoria
- Georgia (2):
  - Site Number - 8002, Tbilisi
  - Site Number - 8000, Tbilisi
- Germany (4):
  - Site Number - 6502, Tübingen, Baden-Wurttemberg
  - Site Number - 6500, Erlangen, Bavaria
  - Site Number - 6501, Oldenburg, Lower Saxony
  - Site Number - 6503, Bochum, North Rhine-Westphalia
- Greece (7):
  - Site Number - 3902, Attiki, Athens
  - Site Number - 3901, Athens, Attica
  - Site Number - 3903, Thessaloniki, Central Macedonia
  - Site Number - 3905, Thessaloniki, Central Macedonia
  - Site Number - 3906, Heraklion, Crete
  - Site Number - 3900, Attiki
  - Site Number - 3904, Larissa
- Poland (7):
  - Site Number - 3004, Poznan, Greater Poland Voivodeship
  - Site Number - 3005, Gorzów Wielkopolski, Lubusz Voivodeship
  - Site Number - 3000, Warsaw, Masovian Voivodeship
  - Site Number - 3001, Warsaw, Masovian Voivodeship
  - Site Number - 3006, Rzeszów, Pakistan
  - Site Number - 3002, Rzeszów, Podkarpackie Voivodeship
  - Site Number - 3003, Lodz
- Puerto Rico (3):
  - Site Number-1029, Caguas
  - Site Number - 1037, Ponce
  - Site Number - 1036, San Juan
- Serbia (3):
  - Site Number - 9000, Belgrade
  - Site Number - 9001, Belgrade
  - Site Number - 9003, Novi Sad
- Spain (6):
  - Site Number - 7104, Badalona, Catalonia
  - Site Number - 7105, Pamplona, Navarre
  - Site Number - 7101, Burjassot, Valencia
  - Site Number - 7100, Madrid
  - Site Number - 7102, Madrid
  - Site Number - 7103, Málaga
- United Kingdom (3):
  - Site Number - 7002, Leeds, West Yorkshire
  - Site Number - 7003, London
  - Site Number - 7000, Manchester

IPD SHARING:
Plan to Share IPD: No